CLINICAL TRIAL: NCT07133880
Title: Differentiating the Effects of Long-acting Bronchodilators Administered by Nebulizer Versus Dry Powder Inhaler in Symptomatic Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Compare the Effects of Nebulizer Versus Inhaler Based Therapy for COPD Using Long-acting Bronchodilators
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Tennessee Graduate School of Medicine (Other)
Collaborators: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4889; Institutional Review Board (Other: The University of Tennessee Health Science Center)
Record Dates: First submitted 2025-08-04; First posted 2025-08-21 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Nebulizer; Dry Powder Inhaler
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — GSK573719; vilanterol; revefenacin; Formoterol Fumarate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DPI Treatment Group (Active Comparator): Group A: Receives Umeclidinium 62.5 µg and Vilanterol 25 µg via DPI and Revefenacin placebo and formoterol placebo (sterile normal saline) via nebulizer at treatment visit # 2 and will continue with assigned treatment and placebo for 12 weeks
  Interventions: Drug: umeclidinium 62.5 µg and vilanterol 25 µg; Drug: Placebo ( Revefenacin and Formoterol )
- Nebulizer Treatment Group (Active Comparator): Group B: Receives revefenacin 175 µg and formoterol 20 µg via nebulizer and placebo DPI at treatment visit # 2 and will continue with assigned treatment and placebo for 12 weeks
  Interventions: Drug: Revefenacin 175 µg, Formoterol 20 µg; Drug: Placebo DPI

INTERVENTIONS:
Drug: umeclidinium 62.5 µg and vilanterol 25 µg — DPI Treatment
  Other Names: Anoro Ellipta
  Arms: DPI Treatment Group
Drug: Revefenacin 175 µg, Formoterol 20 µg — Nebulizer Treatment
  Other Names: Yupelri; Perforomist
  Arms: Nebulizer Treatment Group
Drug: Placebo ( Revefenacin and Formoterol ) — Placebo Nebulizer Treatment
  Other Names: Normal Saline
  Arms: DPI Treatment Group
Drug: Placebo DPI — Placebo DPI Treatment
  Arms: Nebulizer Treatment Group

SUMMARY:
The purpose of this study is to compare the effectiveness of inhaled bronchodilators delivered via nebulizers vs. dry powder inhalers (DPIs) in symptomatic participants with Chronic Obstructive Pulmonary Disease (COPD) who have airflow obstruction (FEV1/FVC ≤ 70%) and show significant air trapping (RV ≥ 120% of predicted).

The investigators hypothesize that, in patients with symptomatic COPD, therapy with a long-acting anti muscarinic agent/long-acting beta agonist (LAMA/LABA) combination administered by nebulizer will improve hyperinflation (increase in inspiratory capacity and reduction in residual volume) and reduce symptoms related to COPD to a greater extent than LAMA/LABA therapy given by a DPI.

The study aims to demonstrate the following:

1. Compare the values of inspiratory capacity (IC) and residual volume (RV) in patients receiving LAMA/LABA by DPI with those receiving LAMA/LABA by nebulizer
2. Compare patient reported outcomes (COPD Assessment Test (CAT score), Baseline/Transition Dyspnea Index (BDI/TDI) and the St. George Respiratory Questionnaire (SGRQ) in symptomatic patients with COPD receiving LAMA/LABA by DPI with those receiving LAMA/LABA by nebulizer

DETAILED DESCRIPTION:
This is a prospective, randomized, parallel group, double dummy, phase four, 13-week clinical trial with 1:1 allocation comparing long-acting anti-muscarinic agent (LAMA; Umeclidinium 62.5 μg once daily) and long acting beta-agonist (LABA; Vilanterol 25 μg once daily) delivered by DPI (Group A), vs a nebulized LAMA/LABA combination (revefenacin 175 μg once daily and formoterol 20 μg twice daily) (Group B) among symptomatic subjects with stable COPD.

The study begins with a screening visit and run-in period. Patients who are eligible and willing to participate will sign informed consent. They will be trained on the use of the DPI and nebulizer, as well as completion of the daily diary (symptom and medication logs) and questionnaires (CAT, BDI/TDI, SGRQ). Vital signs and a physical examination will be performed, and inspiratory flow rate will be determined using the In-Check DIAL. Medications will be adjusted to ensure clinical stability prior to randomization.

Baseline Study Visit 2 occurs within one week of the screening visit. Prior to this visit, participants must not have taken study medication within 48 hours or rescue medication within 6 hours of pulmonary function testing; otherwise, the visit will be rescheduled. At this visit, medical history, current medications, and adverse events are reviewed. Compliance with the daily diary (symptom and medication logs) is assessed, and participants must demonstrate ≥80% completion to continue. Participants complete CAT, BDI, and SGRQ questionnaires, undergo physical examination and vital sign measurement, and perform baseline pulmonary function testing in a plethysmograph. Eligible participants are then randomized 1:1 to receive either active drugs via DPI (Group A) or nebulizer (Group B), with treatment assignments generated using permuted blocks. Group A receives Anoro Ellipta DPI plus nebulized Revefenacin and Formoterol placebos, while Group B receives nebulized Revefenacin and Formoterol plus placebo DPI. The nebulizer is always administered first, followed by the DPI; Time 0 is defined as the end of DPI administration. Post-dose, vital signs and pulmonary function tests are conducted at 1, 2, 4, and 6 hours. Participants also receive training on diary use, study drug/device administration, and medication compliance, and they begin the assigned treatment for 12 weeks with morning and evening doses as per group assignment.

Following Visit 2, patients will continue their assigned treatments twice daily for 12 weeks. Telephone follow-ups will occur at weeks 4 and 8 (Phone Visits 1 and 2) to monitor symptoms, adverse events, and medication adherence, with administration of additional questionnaires.

The final Study Visit 3 will take place at week 12 and will include repeat pulmonary function testing pre-dose and at 1, 2, 4, and 6 hours post-dose, symptom questionnaires, vital signs, and adverse event assessment. Throughout the study, patients will maintain daily symptom diaries, including CAT scores.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 40 years
2. Either sex
3. Current smoker or past cigarette smoking history of > 10 pack-years
4. Symptoms of COPD (cough, sputum production, shortness of breath)
5. Modified Medical Research Council Dyspnea Scale (mMRC) score ≥2 or CAT score ≥10 at Screening/Run-in visit
6. A PIFR > 30 at screening
7. FEV1/FVC ratio < 70% (within the past 12 months)
8. Residual volume (RV) ≥ 120% predicted (within the past 12 months

Exclusion Criteria:

1. Diagnosis of asthma (Verification via medical record and/or patient report)
2. Previously diagnosed atrial fibrillation with rapid ventricular response (heart rate > 110 bpm) or ventricular arrhythmia (ventricular tachycardia) (Verification via medical record and/or patient report)
3. Acute myocardial infarction within 12 weeks of patient study registration (Verification via medical record and/or patient report)
4. Acute exacerbation of congestive heart failure (Verification via medical record and/or patient report)
5. Acute exacerbation of COPD within 8 weeks (Verification via medical record and/or patient report)
6. Recent (within 8 weeks) h/o eye surgery (Verification via medical record and/or patient report)
7. Uncontrolled glaucoma (Verification via medical record and/or patient report)
8. Known diagnosis of liver cirrhosis (Verification via medical record and/or patient report)
9. Known diagnosis of chronic renal insufficiency (defined as a previous serum creatinine > 2.5 mg/dL - Verification via medical record and/or patient report)
10. Intolerance to any of the study drugs
11. Patients receiving long-term azithromycin
12. Planned surgery requiring hospital admission within 3 months
13. Currently enrolled in a pulmonary rehabilitation program
14. Inability to give informed consent
15. Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception (i.e., oral contraceptives, intrauterine devices, diaphragm, or subdermal implants)
16. Inability to understand instructions or comply with the study protocol
17. Participation in another investigational drug clinical trial within 30 days of patient study registration

Medical history can be confirmed by medical records and/or verbal confirmation from patients. However, Inclusion criteria 6 & 7 must be verified by a previous PFT report dated within 6 months of screening

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Difference Between the Values of Area Under the Response Curve for Inspiratory Capacity (IC) | From baseline (Visit 2, Week 2) through study completion (Visit 3, Week 12)
  Difference between the values of area under the response curve for inspiratory capacity (IC) from baseline through six hours (AUC IC 0-6h) after inhalation of LAMA/LABA combination with a nebulizer versus a DPI OR Proportion of participants achieving improvement of >2 points in their CAT score compared to baseline OR Proportion of participants achieving reduction of 4 points in SGRQ score compared to baseline

SECONDARY OUTCOMES:
Percentage change in Residual Volume (RV) from baseline after inhalation of LAMA/LABA combination with a nebulizer versus a DPI | From pre-dose (baseline measurement) to post-dose measurements at 1, 2, 4, and 6 hours during study visit 2 (Week 2) and study visit 3 (Week 12)
Percentage change in Total Lung Capacity (TLC) from baseline after inhalation of LAMA/LABA combination with a nebulizer versus a DPI | From pre-dose (baseline measurement) to post-dose measurements at 1, 2, 4, and 6 hours during study visit 2 (Week 2) and study visit 3 (Week 12)
Percentage change in airway resistance (Raw) from baseline after inhalation of LAMA/LABA combination with a nebulizer versus a DPI | From pre-dose (baseline measurement) to post-dose measurements at 1, 2, 4, and 6 hours during study visit 2 (Week 2) and study visit 3 (Week 12)
Maximum percentage change in inspiratory capacity between 0 and 6 hours after LAMA/LABA combination with a nebulizer versus a DPI | From pre-dose (baseline measurement) to post-dose measurements at 1, 2, 4, and 6 hours during study visit 2 (Week 2) and study visit 3 (Week 12)
Maximum percentage change in RV between 0 and 6 hours after LAMA/LABA combination | From pre-dose (baseline measurement) to post-dose measurements at 1, 2, 4, and 6 hours during study visit 2 (Week 2) and study visit 3 (Week 12)
Maximum Percentage Change in Airway Resistance (Raw) between 0 and 6 hours after LAMA/LABA | From pre-dose (baseline measurement) to post-dose measurements at 1, 2, 4, and 6 hours during study visit 2 (Week 2) and study visit 3 (Week 12)
Correlation of peak inspiratory flow rate with peak IC change from baseline | From pre-dose (baseline measurement) to post-dose measurements at 1, 2, 4, and 6 hours during study visit 2 (Week 2) and study visit 3 (Week 12)
Comparison of CAT scores in patients receiving medications with DPI vs nebulizer | From baseline (Visit 2, Week 2) through study completion (Visit 3, Week 12)
Comparison of SGRQ scores in patients receiving medications with DPI vs nebulizer | At baseline (Visit 2, Week 2), and at study completion (Visit 3, Week 12)
Change in TDI in patients receiving medications with DPI vs nebulizer | Measured at Week 4 (Phone Visit 1), Week 8 (Phone Visit 2), and Week 12 (Study Visit 3)
Change in CAT scores in patients receiving medications with DPI vs nebulizer | From baseline (Visit 2, Week 2) through study completion (Visit 3, Week 12)
Change in SGRQ scores in patients receiving medications with DPI vs nebulizer | Measured at study visit 2 at week 2 and study completion visit 3 at week 12
Correlation of CAT with LF and LH change (inspiratory capacity and residual volume change) with patient-reported outcomes including the SGRQ and the TDI | Baseline (Visit 2) through Study Completion (Visit 3 / Week 12)
Correlation of LH with patient-reported outcomes including scores from the CAT, SGRQ and TDI | Baseline (Visit 2) through Study Completion (Visit 3 / Week 12)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Tennessee Graduate School of Medicine, Knoxville, Tennessee, United States

DOCUMENTS (1):
  • Study Protocol (2024-10-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT07133880/Prot_000.pdf